CLINICAL TRIAL: NCT05586672
Title: High Resolution Electroencephalogram Contribution in Prognostic Evaluation of Language Development in Children With Autism Spectrum Disorder
Brief Title: HR-EEG Contribution in Prognostic Evaluation of Language Development in Children With ASD
Acronym: EE-TSA-LANG
Status: Not yet recruiting | Type: Observational
Sponsor: Etablissement Public de Santé Barthélemy Durand (Other)
Responsible Party: Sponsor
Other Study IDs: 22P01; 2022-A01657-36 (Registry Identifier: ANSM)
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Autism Spectrum Disorder; Language Development; Neurocognitive Disorders; Child Language
Keywords: High Resolution electroencephalogram; Child; Autism Spectrum Disorder; Language
MeSH Terms: conditions — Autism Spectrum Disorder; Neurocognitive Disorders; Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD group: Participants aged from 3 years to 4 years and half at inclusion will be clinically evaluated with standardized scales and tests and will performed an EEG-HR recording while listening to successive soundtracks at several times.
  Interventions: Device: EEG-HR; Diagnostic Test: ADI-R; Diagnostic Test: ADOS-2; Diagnostic Test: IDE; Diagnostic Test: MSEL; Diagnostic Test: Dunn
- Control group: Participants aged from 3 years to 4 years and half at inclusion will be clinically evaluated with standardized scales and tests and will performed an EEG-HR recording while listening to successive soundtracks in inclusion visit.
  Interventions: Device: EEG-HR; Diagnostic Test: ADI-R; Diagnostic Test: ADOS-2; Diagnostic Test: IDE

INTERVENTIONS:
Device: EEG-HR — Passation EEG-HR
Diagnostic Test: ADI-R — Passation of ADI-R scale
  Other Names: AUTISM DIAGNOSTIC INTERVIEW-REVISED
Diagnostic Test: ADOS-2 — Passation of ADOS-2 scale
  Other Names: AUTISM DIAGNOSTIC OBSERVATION SCHEDULE 2
Diagnostic Test: IDE — Passation of IDE scale
  Other Names: Inventaire du Développement de l'Enfant; CDI; Child Development Inventory
Diagnostic Test: MSEL — Passation of MSEL scale
  Other Names: Mullen Scales of Early Learning
  Groups: ASD group
Diagnostic Test: Dunn — Passation of Dunn scale
  Groups: ASD group

SUMMARY:
The goal of this prospective observational multicentric cohort study is to evaluate the clinical prognostic value of the speech tracking score of language development in children with ASD aged from 3 years to 4 years and half at inclusion.

Participants will followed during 4 years with an annual visit. During these visits, each participant will be clinically evaluated (scales and tests) and performed an EEG-HR recording. Two groups will be formed, one with children diagnosed with ASD with language delay, and a control group composed of non-ASD children without language delay, matched on age and gender with the ASD group.

DETAILED DESCRIPTION:
Two groups will be formed, one with children diagnosed with ASD with language delay, and a control group composed of non-ASD children without language delay, matched on age and gender with the ASD group.

- ASD group : For children in the ASD group, 4 visits were planned (inclusion visit, then at one year, two years and three years).

During study visit, each child will be clinically evaluated with standardized scales and tests and will performed an EEG-HR recording while listening to successive soundtracks (modulated pure tones, synthetic voice, recorded voice, real voice, with congruent and non-congruent pictorial supports).

- Control group : For children in the control group, 1 visit was planned : data will be collected at the inclusion visit only.

During this visit, each child will be clinically evaluated with standardized scales and tests and will performed an EEG-HR recording while listening to successive soundtracks (modulated pure tones, synthetic voice, recorded voice, real voice, with congruent and non-congruent pictorial supports).

ELIGIBILITY:
Inclusion Criteria:

For all participants

* Child aged from 3 years to 4 years and half at inclusion.
* Information delivered and no parental objection for study participation.

For ASD group

* Diagnosis of ASD according to DSM-V criteria.
* Expressive language level < 27 months regarding on IDE scale.

For Control group - Matched on age (at +/- 3 months) and gender to ASD group participants.

Exclusion Criteria:

For all participants

* Any illness or treatment that could significantly alter EEG-HR recording (epilepsy, anti-epileptic treatment, psychotropic drugs...).
* Major hearing or vision disorders.

For ASD group

- Severe and characterised neurological pathology other than ASD

For Control group

* Characterised neurological or psychiatric pathology.
* Characteristic language delay.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Child male or female aged from 3 years to 4 years and half at inclusion with ASD or not.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability to discriminate children language development | 4 years
  The primary endpoint is the ability to discriminate children whose language development will be favourable (developmental level ≥ 27 months) from those whose language development will be unfavourable (< 27 months) based on the speech tracking measure (on the EEG-HR at inclusion).

SECONDARY OUTCOMES:
Comparison of speech tracking scores | 4 years
  Comparison of speech tracking scores (phases 1 to 3 of the HR EEG recording protocol).
Evolution of the predictive model | 4 years
  Evolution of the predictive model by integrating data: clinical, longitudinal evolution of speech tracking, deviation from the mean of the control group speech tracking and evolution of speech tracking.
Measures of association by synchronous and diachronic analyses | 4 years
  Measures of association by synchronous and diachronic analyses (mixed generalized linear models for repeated measures).

CONTACTS AND LOCATIONS:
Overall Officials: Mariette Vinurel, Principal Investigator — Etablissement Public de Santé Barthélemy Durand
Locations (1):
- Etablissement Public de Santé Barthélemy Durand, Étampes, France

IPD SHARING:
Plan to Share IPD: No